CLINICAL TRIAL: NCT06275906
Title: Influence of a Different Percentage of Nutrients on the Effects of a Low-calorie Mediterranean Diet Associated With Physical Exercise on the Parameters of Steatosis, Intestinal Function and Metabolic Risk in Patients With Obesity and NAFLD
Brief Title: Influence of a Mediterranean Diet Combined With a Physical Activity Intervention, on NAFLD and Inflammation Parameters.
Acronym: NAFLD-POS5
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Collaborators: Russo Francesco (Unknown); Cozzolongo Raffaele (Unknown); Shahini Endrit (Unknown); Zappimbulso Marianna (Unknown); Giannuzzi Vito (Unknown); De Nucci Sara (Unknown); Rinaldi Roberta (Unknown); Sila Annamaria (Unknown); Tatoli Rossella (Unknown); Cerabino Nicole (Unknown); Donghia Rossella (Unknown); Franco Isabella (Unknown); Bianco Antonella (Unknown); Curci Ritanna (Unknown); Bagnato Claudia Beatrice (Unknown); Sciarra Sabrina (Unknown); Prospero Laura (Unknown); Serino Grazia (Unknown); Scalavino Viviana (Unknown); Piccinno Emanuele (Unknown); Pesole Pasqua Letizia (Unknown); Coletta Sergio (Unknown); Stabile Dolores (Unknown); Riezzo Giuseppe (Unknown); Ancona Anna (Unknown); D'Attoma Benedetta (Unknown); Ignazzi Antonia (Unknown)
Responsible Party: Principal Investigator, Prof. Giovanni De Pergola, MD, Prof., MD, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NAFLD-POS5
Record Dates: First submitted 2024-02-05; First posted 2024-02-23 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: NAFLD; Obesity; IBS
Keywords: NAFLD; Obesity; Mediterranean diet; physical activity; walk
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity; Motor Activity | interventions — Diet, Mediterranean

STUDY DESIGN:
Intervention Model Description: The study evaluates the effects of two different Mediterranean Diet models, based on different percentages of macronutrients, on NAFLD and Metabolic Risk.
  The Mediterranean Diet is associated with a program of moderate intensity aerobic physical exercise (walking) carried out 3 times a week for 3 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm 1 (Experimental): The 1st arm involves a low-calorie diet, which respects the criteria of the Mediterranean diet, with the following macronutrient percentage: carbohydrates 50% of total calories, lipids 30% of total calories, proteins 20% of total calories.
  The dietary intervention will be combined with moderate intensity exercise (outdoor walking).
  Interventions: Other: Mediterranean diet and moderate intensity physical exercise (outdoor walking).
- Intervention arm 2 (Experimental): The 2nd arm involves a low-calorie diet, which respects the criteria of the Mediterranean diet, with the following percentage of macronutrients: carbohydrates 30% of total calories, lipids 50% of total calories, proteins 20% of total calories.
  The dietary intervention will be combined with moderate intensity exercise (outdoor walking).
  Interventions: Other: Mediterranean diet and moderate intensity physical exercise (outdoor walking).

INTERVENTIONS:
Other: Mediterranean diet and moderate intensity physical exercise (outdoor walking). — Mediterranean Diet, based on the different percentage of carbohydrates and lipids, associated with a program of moderate intensity aerobic physical exercise (outdoor walking), in patients with obesity and NAFLD.

SUMMARY:
The study in question is an interventional study with nutritional intervention.

The aim of the study is to evaluate whether the adoption of two different models of Mediterranean Diet, based on the different percentage of carbohydrates and lipids, associated with a program of moderate intensity aerobic physical exercise, in patients with obesity and NAFLD can exercise, after only 3 months, effects on:

* specific aspects associated with NAFLD, such as the degree of hepatic steatosis and fibrosis;
* circulating levels of molecules correlated with the degree of generalized and hepatic inflammation and the blood concentrations of metabolic and cardiovascular risk factors associated with abdominal obesity;
* intestinal barrier;
* body composition;
* intestinal microbiota;
* symptoms of IBS (irritable bowel syndrome) in patients with NAFLD.

DETAILED DESCRIPTION:
BACKGROUND Chronic liver diseases are among the main causes of morbidity and mortality. Increasing liver disease mortality has been associated with increasing prevalence of NAFLD. The term "fatty liver disease" is the hallmark of NAFLD and refers to a fat deposit in liver cells greater than 5% that is not related to alcohol intake, viral infections, or drug use. Hepatic steatosis is an independent risk factor for all liver alterations that characterize NAFLD and, in particular, inflammation and fibrosis.

The percentage of NAFLD tends to increase with increasing BMI, Age, Presence of metabolic diseases such as dyslipidemia, Type 2 diabetes.

The following are involved in the onset and progression of NAFLD:

* insulin resistance
* generalized inflammation;
* intestine-liver pathways
* intestinal microbiota. In the absence of officially approved pharmacological therapies for the treatment of NAFLD, the guidelines recommend lifestyle-based interventions, both in quantitative and qualitative terms in diet and increased physical exercise. Diet can improve NAFLD by reducing the amount of liver fat and insulin resistance, while exercise promotes weight loss and improves liver function.

Limiting calorie intake in diets, reducing alcohol consumption, and reducing consumption of highly processed foods have proven to be the most important factor in the management of NAFLD.

Regarding the Mediterranean diet, although there are studies demonstrating its effectiveness in improving NAFLD, there are no publications that have examined which Mediterranean diet model is best for NAFLD with regards to macronutrient content. In the Mediterranean diet, carbohydrates are mainly supplied by foods rich in fiber and with a low glycemic index or low glycemic load, while lipids are mainly supplied by foods rich in monounsaturated fatty acids (mainly olive oil) and polyunsaturated fatty acids (mainly dried fruit, fish and vegetables). It is not known whether variations in the proportion of carbohydrates and lipids, which characterize the Mediterranean diet, can favorably or unfavorably influence the development of NAFLD and NASH.

It has been shown that physical exercise, reduces the amount of liver fat and this change is associated with changes in body weight and cardiorespiratory capacity.

Recent studies suggest that changes in the gut microbiota may represent a new strategy to prevent or treat NAFLD.

A recent prospective study observed that NAFLD is associated with a 20% increased risk of developing irritable bowel syndrome (IBS), a disease characterized by abdominal pain and bloating, frequent diarrhea or prolonged constipation, often alternating periodic.

Since NAFLD and IBS share changes in circulating levels of proinflammatory cytokines, increased (TNF)-α, interleukin (IL)-6, and decreased IL-10, alterations in the intestinal barrier, and alterations in intestinal motility, one cannot exclude that improvement or worsening of NFLD could influence improvement or worsening of IBS.

Inflammation associated with obesity may in turn play a significant role in the development of gastrointestinal disorders. It is a chronic state of low intensity that involves the entire organism. Obesity is related to an increase in inflammatory cytokines in tissues that activate immune responses, altering cellular metabolic pathways. Chronic low intensity inflammation and the variation in the concentration of metabolic hormones, together with the distribution of adipose tissue in the abdominal cavity and alterations in the bacterial populations of the intestinal microbiota, represent the main factors involved in the development of gastrointestinal diseases. Pathologies that develop precisely through alterations of the intestinal barrier. When evaluating the integrity of the intestinal barrier, it is important to consider zonulin, a GI peptide capable of modulating the functionality of tight junctions.

Serum zonulin levels have been shown to correlate with the extent of damage to the mucosal barrier. Cellular and/or TJ damage can impact proper leaky gut function. I-FABPs are cytosolic proteins present in epithelial cells responsible for the transport of fatty acids and are released into circulation following the loss of membrane integrity and eliminated in the urine and represent a non-invasive marker of damage at the epithelial level intestinal.

Alterations in the barrier function can favor the entry of bacteria and their products. Lipopolysaccharide (LPS) has been found to influence barrier function. Under physiological conditions, LPS is unable to cross intact epithelium, but in the presence of reduced epithelial integrity it is able to cross the gastrointestinal barrier.

Tryptophan, an essential amino acid for humans, is catabolized by commensal bacteria into various derivatives, which are absorbed by the intestine and eliminated in the urine. Two of these compounds, indole and skatole, are currently used to diagnose dysbiosis of the small intestine and colon, respectively.

CLINICAL STUDY DESIGN The study, conducted on patients with both obesity (BMI > 30.0) and NAFLD (diagnosed by FLI (fatty liver index) and/or Fibroscan will be a two-arm interventional study, with nutritional and increased physical exercise. The enrolled patients, who meet the inclusion criteria, will be randomly assigned to one of the two study arms and will be asked to follow a personalized diet based on anthropometric characteristics, following the percentage of macronutrients in their arm. All patients will be asked to follow a low-calorie diet, with ¾ of the calories of an isocaloric diet. The exercise program administered to patients will be the same for everyone. Having established common criteria for patient recruitment (presence of obesity and NAFLD), type of low-calorie diet (3/4 of an isocaloric diet) and type of physical exercise, patients will be enrolled and randomly assigned to the two intervention arms. Arm 1 involves a low-calorie diet, meeting the criteria of the Mediterranean diet, with the following percentage of macronutrients: carbohydrates 50% of total calories, lipids 30%, proteins 20%; Arm 2 involves a low-calorie diet, meeting the criteria of the Mediterranean diet, with the following percentage of macronutrients: carbohydrates 30% of total calories, lipids 50%, proteins 20%.

The exercise will be structured and organised. An effective prescription includes an exercise program that is systematically designed and personalized in terms of frequency, intensity, time, type, volume and progression.

Frequency. Physical activity (walking) will be carried out outdoors on an urban route 3 times a week, on non-consecutive days, for 12 weeks.

Intensity. The intensity of the exercise (50/75% of max HR) Type. The type of exercise is moderate aerobic with a speed ranging from 5 to 10 km/h.

Time. Outing lasting 60 minutes The treatment will last 3 months and, in addition to the V0 (Screening Visit), a further 3 visits are planned (V1-V2-V3).

Patients with obesity (BMI > 30.0) and NAFLD, who are not stably taking drugs, will be considered potentially eligible for enrollment.

At V0 potentially enrollable patients, will undergo:

* Anamnesis;
* Fibroscan, to assess the degree of hepatic steatosis;
* Survey of anthropometric characteristics
* Bioimpedance examination;
* Body composition assessment by DEXA
* Delivery of the accelerometer to the patient, on loan for use for the next 7 days.
* Completion of IPAQ-SF and sports history. If the inclusion criteria are met, the enrolled patients will be invited to return for V1, after 7 days to receive the dietary plan and will be asked to complete two questionnaires assessing gastrointestinal symptoms, Irritable Bowel Syndrome - Severity Scoring System (IBS-SSS), specific to IBS symptoms, and Gastrointestinal Symptom Rating Scale (GSRS), which evaluates gastrointestinal symptoms more generally. Patients will also be asked to complete the Morningness-Eveningness Questionnaire (MEQ-SA). Intestinal characteristics will be assessed using the Bristol scale before, during and after the intervention period.

At V1 patients will also undergo a blood sample via venipuncture. They will be asked to bring two stool samples for the evaluation of intestinal microbiota, fecal zonulin and fecal metabolome. You will also be asked to bring two urine samples. Stool and urine samples will be requested for each visit (V1-V2-V3) Microbiome characterization will be performed using a DNA metabarcoding and metatranscriptomics approach. DNA metabarcoding analysis will be conducted using the V5-V6 hypervariable regions of 16S rRNA for bacteria (MiSeq-Illumina platform). The samples found to be significant in the DNA metabarcoding analysis will be subjected to metatracryptomic analysis (NextSeq 500 platform - Illumina). Metagenomic and metatracryptomic data will be analyzed using bioinformatics pipelines.

Metabolomics examinations will be performed on stool and urine samples. Barrier peptide assay: assays of faecal and serum Zonulin, as well as I-FABP, DAO and circulating LPS in serum will be performed using commercially available ELISA methods.

Dosage of indole and skatole in urine: indole is dosed with a colorimetric analytical method while skatole is determined with a chromatographic method with fluorometric detection on urine collected early in the morning. When urinary indole and skatole values exceed the normal threshold they express fermentative (in the small intestine) and putrefactive (in the colon) dysbiosis respectively.

During V1 patients will also be given a GI Symptom Diary to fill in until the next visit, as well as for subsequent visits.

Additionally there will be:

* Muscle strength measurement test: HandGripp test;
* Test for measuring physical performance: SPPB;
* Dynamic balance test: (TGUG, Time Get Up and Go test)
* 2 km walking test.
* Sit and Reach Test Finally, four questionnaires will be administered to assess levels of anxiety, depression and stress. Specifically, the Hospital Anxiety and Depression Scale (HADS) and Perceived Stress Scale (PSS), the Rotter Locus of Control Scale (Q_LOC), and the Delaying Gratification Inventory (DGI).

Patients will be recalled after 45 days (V2) and 90 days (V3).

During these visits they will be subjected to:

* blood sampling by venipuncture;
* GSRS questionnaire;
* IBS-SSS questionnaire;
* Detection of anthropometric characteristics;
* Bioimpedance test

In V3 alone, patients will also undergo:

* Completion of the HADS questionnaire (Hospital Anxiety and Depression Scale);
* Completion of the PSS (Perceived Stress Scale) questionnaire;
* Completion of Rotter's locus of control scale (Q_LOC) questionnaire
* Completion of the Delaying Gratification Inventory (DGI) questionnaire.
* Test for measuring muscle strength HandGripp Test;
* Test for measuring physical performance: SPPB;
* Dynamic balance test: (TGUG, Time Get Up and Go test)
* 2-Km Walking Test.
* Sit and Reach Test The blood sample taken at the V1-V2-V3 examinations will be used for the dosage of routine haematochemical parameters and nutritional, metabolic and cardiovascular risk parameters (Glycaemia, insulin glycated haemoglobin, triglycerides, total cholesterol, HDL and LDL cholesterol, transaminases (AST and ALT), γGT, creatininemia, uricinemia, blood count, ferritin, 25-OH-vitamin D, calcemia, IGF-I, TSH, FT3, FT4, proBNP). Based on the results, the degree of insulin resistance (HOMA index) and the degree of hepatic steatosis FLI, (fatty liver index) will be calculated, based on anthropometric (BMI, abdominal circumference) and haematochemical (triglycerides and γGT) parameters.) and liver fibrosis (FIB-4).

Major adipokines (leptin, adiponcetin, RBP-4, resistin, visfatin, chemerin), major hepatic growth factors (HGF, Fetuin-A, FGF21, FGF19, PAI-1), major pro-inflammatory cytokines (high-sensitivity C-reactive protein, IL-6, IL-8 and TNF-α) and anti-inflammatory cytokines (IL-4) will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 30 Kg/m2 or an abdominal circumference (waist) > 94 cm in men and > 80 cm in women (IDF criteria for the definition of abdominal obesity) with or without the characteristics that characterize metabolic syndrome
* Age range between 18 and 60 years, both sexes
* Diagnosis of hepatic steatosis, formulated on the basis of recognized criteria (fibroscan [CAP (controlled attenuation parameter) > 238 dB/m], FLI).

Exclusion Criteria:

* Normal weight and underweight subjects
* Presence of any pathology that could influence the presence of steatosis apart from the pathologies that represent inclusion criteria
* Treatment with any device, pharmacological or otherwise, which can influence hepatic metabolism and, therefore, the presence of steatosis
* Pregnancy or breastfeeding
* Subjects with osteo-articular pathologies that may prevent regular physical exercise

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2025-04-08 (Estimated); Study Completion 2026-04-08 (Estimated)

PRIMARY OUTCOMES:
The effect of intervention on CAP value | at Baseline and after 90 days
  To evaluate whether the adoption of one of the two different models of the Mediterranean diet, based on different percentages of carbohydrates and lipids, combined with a moderate-intensity aerobic exercise programme, in patients with obesity and NAFLD can exert favourable effects on the CAP value and the degree of liver fibrosis assessed by Fibroscan after only 3 months.
  Values considered normal are less than 5.1 kPa (kPascal)
The effect of intervention on FLI value | at Baseline and after 90 days
  To evaluate whether the adoption of one of the two different models of the Mediterranean diet, based on different percentages of carbohydrates and lipids, combined with a moderate-intensity aerobic exercise programme, in patients with obesity and NAFLD can exert favourable effects on the FLI value (fatty liver index), based on anthropometric parameters (BMI, abdominal circumference) and blood chemistry (triglycerides and γGT).
  Values considered normal are less than 30.
The effect of intervention on routine blood chemistry parameters, relating to NAFLD and fibrosis, nutritional status, inflammatory status and metabolic and cardiovascular risk | at Baseline and after 90 days
  To evaluate whether the adoption of one of two different Mediterranean diet models, based on different percentages of carbohydrates and lipids, combined with a moderate intensity aerobic exercise program, in patients with obesity and NAFLD can exert favorable effects on routine blood chemistry tests parameters, relating to NAFLD, fibrosis, nutritional and inflammatory status, metabolic and cardiovascular risk.
  The following will be considered: blood sugar, insulin, glycated hemoglobin, triglycerides, total cholesterol, HDL and LDL, transaminases, γGT, creatinine, uric acid, blood count, ferritin, vitamin D, calcemia, IGF-I, TSH, FT3, FT4, proBNP and HOMA INDEX, adipokines (leptin, adiponcetin, RBP-4, resistin, visfatin, chemerin), hepatic growth factors (HGF, Fetuin-A, FGF21, FGF19, PAI-1) and proinflammatory cytokines (C-Reactive Protein, IL-6, IL-8, TNF-α) and anti-inflammatory (IL-4).
The effect of the intervention on the integrity of the intestinal barrier | at Baseline and after 90 days
  To evaluate whether the adoption of one of two different Mediterranean diet models, based on different percentages of carbohydrates and lipids, combined with a moderate intensity aerobic exercise program, in patients with obesity and NAFLD can exert favorable effects on the function and integrity of the intestinal barrier assessed by measuring Zonulin, I-FABP, DAO.

SECONDARY OUTCOMES:
The effect of the intervention on the Gastrointestinal Symptoms | at Baseline and after 90 days
  To evaluate whether the adoption of one of the two different models of the Mediterranean diet, based on different percentages of carbohydrates and lipids, combined with a moderate-intensity aerobic exercise programme, in patients with obesity and NAFLD can exert favourable effects on the GI symptoms (IBS or functional dyspepsia or functional bloating)
The effect of the intervention on the Body Composition | at Baseline and after 90 days
  To evaluate whether the adoption of one of two different Mediterranean diet models, based on different percentages of carbohydrates and lipids, combined with a moderate intensity aerobic exercise program, in patients with obesity and NAFLD can exert favorable effects on body composition measured by BIA and anthropometric parameters.

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Saverio de Bellis, Castellana Grotte, BARI, Italy

REFERENCES:
- [Background] Younossi ZM, Golabi P, Paik JM, Henry A, Van Dongen C, Henry L. The global epidemiology of nonalcoholic fatty liver disease (NAFLD) and nonalcoholic steatohepatitis (NASH): a systematic review. Hepatology. 2023 Apr 1;77(4):1335-1347. doi: 10.1097/HEP.0000000000000004. Epub 2023 Jan 3. PMID 36626630
- [Background] Younossi Z, Anstee QM, Marietti M, Hardy T, Henry L, Eslam M, George J, Bugianesi E. Global burden of NAFLD and NASH: trends, predictions, risk factors and prevention. Nat Rev Gastroenterol Hepatol. 2018 Jan;15(1):11-20. doi: 10.1038/nrgastro.2017.109. Epub 2017 Sep 20. PMID 28930295
- [Background] Haigh L, Kirk C, El Gendy K, Gallacher J, Errington L, Mathers JC, Anstee QM. The effectiveness and acceptability of Mediterranean diet and calorie restriction in non-alcoholic fatty liver disease (NAFLD): A systematic review and meta-analysis. Clin Nutr. 2022 Sep;41(9):1913-1931. doi: 10.1016/j.clnu.2022.06.037. Epub 2022 Jul 2. PMID 35947894
- [Background] Baker CJ, Martinez-Huenchullan SF, D'Souza M, Xu Y, Li M, Bi Y, Johnson NA, Twigg SM. Effect of exercise on hepatic steatosis: Are benefits seen without dietary intervention? A systematic review and meta-analysis. J Diabetes. 2021 Jan;13(1):63-77. doi: 10.1111/1753-0407.13086. Epub 2020 Aug 11. PMID 32667128
- [Background] Wu S, Yuan C, Yang Z, Liu S, Zhang Q, Zhang S, Zhu S. Non-alcoholic fatty liver is associated with increased risk of irritable bowel syndrome: a prospective cohort study. BMC Med. 2022 Aug 22;20(1):262. doi: 10.1186/s12916-022-02460-8. PMID 35989356
- [Background] Kawaguchi T, Takahashi H, Gerber LH. Clinics in Liver Disease: Update on Nonalcoholic Steatohepatitis: Sarcopenia and Nonalcoholic Fatty Liver Disease. Clin Liver Dis. 2023 May;27(2):275-286. doi: 10.1016/j.cld.2023.01.005. Epub 2023 Feb 26. PMID 37024207
- [Background] Martin-Rincon M, Perez-Valera M, Morales-Alamo D, Perez-Suarez I, Dorado C, Gonzalez-Henriquez JJ, Juan-Habib JW, Quintana-Garcia C, Galvan-Alvarez V, Pedrianes-Martin PB, Acosta C, Curtelin D, Calbet JAL, de Pablos-Velasco P. Resting Energy Expenditure and Body Composition in Overweight Men and Women Living in a Temperate Climate. J Clin Med. 2020 Jan 11;9(1):203. doi: 10.3390/jcm9010203. PMID 31940840